CLINICAL TRIAL: NCT04672798
Title: The Center for Enhancing Treatment & Utilization for Depression and Emergent Suicidality Phase 2-Study 3-BRITEPath
Brief Title: BRITEPath- Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Stepp, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY20110359; P50MH115838-02 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Depression; Suicidal Ideation
Keywords: depression; suicidal ideation; anxiety; treatment; app; safety planning; provider
MeSH Terms: conditions — Depression; Suicidal Ideation; Anxiety Disorders; Alzheimer Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study will use a parallel study design, where participants are randomized into two groups, BRITEPath or TAU, and will receive interventions in parallel.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRITEPath (Experimental): Participants will receive the components in BRITEPath from a mental health (MH) clinical trained by the study staff/PI's on how to implement BRITE safety planning with fidelity.
  First, the MH clinician will review possible barriers to implementation of the safety plan and problem-solve appropriately with patient and parent(s); (2) BRITE is the emotion regulation/safety planning app loaded on the patient's smartphone that populated with support from Guide2BRITE; and (3) BRITEBoard, a clinician dashboard that shows app use, change in distress and symptoms ratings, and can be used for shared decision making with parents, patients, and PCPs. Clinicians will review adolescent's skill development and app content with parents. Prior to discharge or following acute increases in suicide risk.
  Interventions: Behavioral: BRITEPath
- Treatment As Usual (TAU) (Active Comparator): Participants in the TAU group will receive treatment from their mental health clinician which may include safety planning.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: BRITEPath — BRITEPath will guide co-located mental health clinicians in the use of an emotion regulation and safety planning app (BRITE) to be loaded on the phone of depressed and suicidal adolescents in order to improve depression and reduce the likelihood of a suicide attempt.
  Arms: BRITEPath
Behavioral: Treatment As Usual (TAU) — Participants in this group will receive usual care from their mental health care provider.
  Arms: Treatment As Usual (TAU)

SUMMARY:
BRITEPath (BP) aims to support co-located mental health clinicians in the development of a high quality, effective, and personalized safety plan for referred patients who screen positive for depression and/or suicidal ideation.

BRITEPath utilizes BRITE, a safety planning and emotion regulation app that is loaded on the patient's smart phone and has previously been shown to be well accepted and to reduce suicide attempts compared to usual care in psychiatric inpatients (HR = 0.49). To support mental health clinicians in the development of effective safety plans, study investigators will develop Guide2Brite (G2B), which provides step-by-step instructions for the mental health clinician on how to populate BRITE onto the patient's smartphone and BRITEBoard, a clinician dashboard that tracks patient symptoms, app use, and rating on helpfulness of different interventions assessed through BRITE.

DETAILED DESCRIPTION:
BRITEPath has 3 components: 1) BRITE, an emotion regulation and safety planning phone app that is delivered by a co-located mental health (MH) clinician to adolescents at the time of their first therapy appointment; 2) Guide2Brite, which will guide the co-located MH clinician in working with the adolescent to population content onto BRITE; and 3) BRITEBoard, which is a clinician dashboard delivered to the MH clinician and PCP.

Assignment of Interventions: This study will utilize a 1:1 randomization scheme to randomize participants to receive BRITEPath intervention or Treatment as Usual (TAU).

Hypothesis: The use of BRITEPath will decrease depressive symptoms, distress, and suicidality (any self-injurious ideation, urges, or behavior) as well as improve overall functioning compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

1. Youth aged 12-26yo
2. Own a device (e.g. smartphone, iPod, tablet) with capability to download BRITE app
3. Biological or adoptive parent is willing to provide informed consent for teen to participate
4. Youth speaks and understands English
5. Positive PHQ score or provider determines youth has depressive symptoms based on clinical interaction and refers youth to the study (in cases when PHQ is not available and study staff will complete the PHQ during the screening) OR Provider can refer if they are unclear if symptoms are depressive and PHQ scoring will be used to determine youth's eligibility. OR Screening Wizard screening questionnaire (which includes the PHQ and depressive symptom questions) indicates depression OR provider/parent have concern that youth/patient has a mood or behavioral problem
6. Family agrees to see an (embedded) MH therapist at the practice
7. PHQ scores: Score of 8 or higher on PHQ-8 -or- Score of 1 or higher on #9 of PHQ-9 suicidality item

Exclusion Criteria:

1. Non English speaking
2. No parent willing to provide informed consent
3. No cell phone capability of downloading BRITE app
4. Is currently experiencing mania or psychosis
5. Evidence of an intellectual or developmental disorder (IDD)
6. Life threatening medical condition that requires immediate treatment (including emergent suicidality, homicidally, abuse/neglect, or other mental or physical condition)
7. Other cognitive or medical condition preventing youth from understanding study and/or participating.
8. Currently receiving MH treatment/currently satisfied with treatment

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Stepp, PhD, Principal Investigator — University of Pittsburgh; David Brent, MD, Study Director — University of Pittsburgh
Locations (6):
- United States (6):
  - Henry Ford Health System, Detroit, Michigan
  - Northwell Hospital, Hyde Park, New York
  - Children's Community Pediatrics (CCP-Moon) of Children's Hospital of Pittsburgh of UPMC, Moon Township, Pennsylvania
  - STAR- Center, Pittsburgh, Pennsylvania
  - Children's Community Pediatrics (CCP- Wexford) of Children's Hospital of Pittsburgh of UPMC, Wexford, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

RESULTS

PARTICIPANT FLOW:
Groups:
- BRITEPath: Participants will receive the components in BRITEPath from a mental health (MH) clinical trained by the study staff/PI's on how to implement BRITE safety planning with fidelity.
  First, the MH clinician will review possible barriers to implementation of the safety plan and problem-solve appropriately with patient and parent(s); (2) BRITE is the emotion regulation/safety planning app loaded on the patient's smartphone that populated with support from Guide2BRITE; and (3) BRITEBoard, a clinician dashboard that shows app use, change in distress and symptoms ratings, and can be used for shared decision making with parents, patients, and PCPs. Clinicians will review adolescent's skill development and app content with parents. Prior to discharge or following acute increases in suicide risk.
  BRITEPath: BRITEPath will guide co-located mental health clinicians in the use of an emotion regulation and safety planning app (BRITE) to be loaded on the phone of depressed and suicidal adolescents in order to improve depression and reduce the likelihood of a suicide attempt.
Period: Overall Study
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Started | 68 | 33
Completed | 59 | 31
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Population: 1 intervention participant did not complete the entire Baseline assessment following consent and PHQ-9 assessment. A total of 67 intervention participants completed all Baseline measures. All 33 TAU participants completed all Baseline assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | BRITEPath | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 68 | 33 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 12 | 42
  Between 18 and 65 years | 38 | 21 | 59
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 15 | 4 | 19
  Female | 43 | 24 | 67
  Female to Male Transgender | 2 | 0 | 2
  Non-binary/ Queer | 8 | 4 | 12
  Other Gender | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 63 | 30 | 93
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 45 | 26 | 71
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 68 | 33 | 101
Depression Severity [Mean (Standard Deviation); unit: score on a scale] — Total scores from the Patient Health Questionnaire (PHQ-9) assesses depression severity. The PHQ-9 is 9 items with scoring ranging from 0-27. The higher the score, the more severe the depression symptoms are. A score of 0-4=no depression; 5-9=mild depression; 10-14=moderate depression; 15-19=moderately severe depression; 20-27=severe depression symptoms. PHQ collected at recruitment for eligibility, baseline, and follow up timepoints to track changes in depression severity over course of study.
  score on a scale | 10.6 (5.9) | 11.4 (5.7) | 10.9 (5.9)
Quality of life and Social/Emotional Functioning [Mean (Standard Deviation); unit: score on a scale] — Pediatric Quality of Life Inventory Version 4 assesses quality of life and functioning. Items on the Pediatric Quality of Life Generic Core Scales are reverse scored & transformed to 0-100 scale. Higher scores indicate better health related quality of life. 0 ("Never") = 100; 1 ("Almost Never") = 75; 2 ("Sometimes") = 50; 3 ("Often") = 25; 4 ("Almost Always") = 0. The total score is Sum of all items over number of items answered. Population: The PEDS QOL measure is only administered to adolescents in the study, not those age 18+. There were young adult participants included in the study in each treatment arm.
  score on a scale
    PEDS QOL Physical Score: number analyzed (Participants) | 21 | 10 | 31
    PEDS QOL Physical Score | 81.7 (20) | 70.5 (18) | 78.1 (19.8)
    PEDS QOL Emotional Score: number analyzed (Participants) | 21 | 10 | 31
    PEDS QOL Emotional Score | 59 (27.1) | 50 (18.4) | 56.1 (24.7)
    PEDS QOL Social Score: number analyzed (Participants) | 21 | 10 | 31
    PEDS QOL Social Score | 77.4 (23.7) | 69.8 (27.9) | 74.9 (25)
    PEDS QOL Psychosocial Health Summary Score: number analyzed (Participants) | 21 | 10 | 31
    PEDS QOL Psychosocial Health Summary Score | 66.6 (22.9) | 56.9 (13.8) | 63.5 (20.7)
    PEDS QOL Total Score: number analyzed (Participants) | 21 | 10 | 31
    PEDS QOL Total Score | 71.8 (20.4) | 61.6 (14.6) | 68.5 (19.1)
Suicidal Ideation and Behavior [Mean (Standard Deviation); unit: score on a scale] — Suicidal attempt & ideation measured through Columbia Suicide Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9). Assign score of 0 if no ideation/behavior present, assign a score of 1 if ideation/behavior present. "Yes" to question 9 (score=1) on PHQ-9 indicates suicidal ideation. "Yes" to suicidal behavior questions (Categories 7-10): 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide indicates respondent has suicidal behavior. Any score greater than 0 is important/may indicate need for intervention. Population: 1 participant only completed demographics and PHQ-9 measure at Baseline after completed consent.
  score on a scale
    PHQ-9-question #9 | 0.5 (0.8) | 0.4 (0.8) | 0.5 (0.8)
    C-SSRS Category 7: Aborted Attempts: number analyzed (Participants) | 67 | 33 | 100
    C-SSRS Category 7: Aborted Attempts | 0 (0.2) | 0 (0) | 0.0 (0.2)
    C-SSRS Category 8: Interrupted Attempts: number analyzed (Participants) | 67 | 33 | 100
    C-SSRS Category 8: Interrupted Attempts | 0 (0.1) | 0 (0.2) | 0.0 (0.1)
    C-SSRS Category 9: Actual Attempts (non-lethal): number analyzed (Participants) | 67 | 33 | 100
    C-SSRS Category 9: Actual Attempts (non-lethal) | 0.1 (0.3) | 0 (0) | 0.1 (0.3)
    C-SSRS Category 10: Completed Suicide: number analyzed (Participants) | 67 | 33 | 100
    C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0) | 0.0 (0.0)
Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication) [Count of Participants; unit: Participants] — The Child and Adolescent Service Assessment (CASA) collects service utilization of all participants to determine the amount of services accessed. The CASA response data displayed are those who responded positively that they received the service. Those who said yes to receiving the service is scored as a 1. Multiple participants can say yes to more than 1 service. Population: 1 participant only completed demographics and PHQ-9 measure at Baseline after completed consent.
  Participants
    Use of Outpatient Services: number analyzed (Participants) | 67 | 33 | 100
    Use of Outpatient Services | 61 | 29 | 90
    Use of School Services: number analyzed (Participants) | 67 | 33 | 100
    Use of School Services | 36 | 20 | 56
    Use of Emergency Services: number analyzed (Participants) | 67 | 33 | 100
    Use of Emergency Services | 11 | 3 | 14
    Use of Legal Services: number analyzed (Participants) | 67 | 33 | 100
    Use of Legal Services | 0 | 1 | 1
    Use of Inpatient Services: number analyzed (Participants) | 67 | 33 | 100
    Use of Inpatient Services | 18 | 7 | 25
    Use of Medications: number analyzed (Participants) | 67 | 33 | 100
    Use of Medications | 57 | 26 | 83

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Total scores from the Patient Health Questionnaire (PHQ-9) will be used to assess depression severity, as a primary outcome. The PHQ-9 is a 9 items assessment with scoring ranging from 0-27. The higher the score, the more severe the depression symptoms are. A score of 0-4= no depression; 5-9= mild depression; 10-14= moderate depression; 15-19= moderately severe depression; 20-27= severe depression symptoms.
Time Frame: At 4 week follow up after Baseline
Population: 6 intervention participants and 1 TAU participant did not complete the PHQ-9 and remain in the "intention to treat" analysis sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 62 | 32
score on a scale | 8.6 (5.6) | 10.8 (5.4)

2. Primary Outcome: Depression Severity
Description: as for outcome 1
Time Frame: At 12 week follow up after Baseline
Population: 9 intervention participants and 2 TAU participants did not complete the PHQ-9 and remain in the "intention to treat" analysis sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 59 | 31
score on a scale | 8.3 (5.4) | 10 (5.9)

3. Primary Outcome: Suicidal Ideation and Behavior
Description: Suicide attempt & ideation is measured through Columbia Suicide Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9). Assign score of 0 if no ideation/behavior present or answer is "No", assign a score of 1 if ideation/behavior present or "Yes." A "Yes" to question 9 (score=1) on PHQ-9 indicates suicidal ideation. Suicidal ideation or behavior= "yes" answer to any of suicidal behavior questions (Categories 7-10) on the CSSRS. 7- Aborted Attempt 8- Interrupted Attempt 9- Actual Attempt (non-fatal) 10- Completed Suicide. Any score greater than 0 is important/may indicate need for intervention and may indicate worse outcomes.
Time Frame: At 4 week follow up after Baseline
Population: 6 intervention participants and 1 TAU participant did not complete the C-SSRS and remain in the "intention to treat" analysis sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 62 | 32
score on a scale
  PHQ-9 question #9 | 0.3 (0.7) | 0.5 (0.9)
  C-SSRS Category 7: Aborted Attempt | 0 (0) | 0 (0)
  C-SSRS Category 8: Interrupted Attempt | 0 (0) | 0 (0)
  C-SSRS Category 9: Actual Attempt (non-fatal) | 0 (0) | 0 (0)
  C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0)

4. Primary Outcome: Suicidal Ideation and Behavior
Description: as for outcome 3
Time Frame: At 12 week follow up after Baseline
Population: 9 intervention participants and 2 TAU participants did not complete the C-SSRS and remain in the "intention to treat" analysis sample
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 59 | 31
score on a scale
  PHQ-9 Question 9 (ideation) | 0.2 (0.5) | 0.4 (0.7)
  C-SSRS Category 7: Aborted Attempt | 0 (0.2) | 0 (0)
  C-SSRS Category 8: Interrupted Attempt | 0 (0) | 0 (0)
  C-SSRS Category 9: Actual Attempt (non-fatal) | 0 (0) | 0 (0)
  C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0)

5. Primary Outcome: Quality of Life and Social/Emotional Functioning
Description: Pediatric Quality of Life Inventory Version 4 assesses quality of life and functioning. Items on the Pediatric Quality of Life Generic Core Scales are reverse scored & transformed to 0-100 scale. Higher scores indicate better health related quality of life. 0 ("Never") = 100; 1 ("Almost Never") = 75; 2 ("Sometimes") = 50; 3 ("Often") = 25; 4 ("Almost Always") = 0. The total score is Sum of all items over number of items answered.
Time Frame: At 4 week follow up after Baseline
Population: Only adolescents under age 18 received the PEDS-QOL measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 19 | 9
score on a scale
  PEDS QOL Physical Score | 89.3 (11.5) | 71.5 (22.5)
  PEDS QOL Emotional Score | 68.7 (25.9) | 60.6 (20.8)
  PEDS QOL Social Score | 81.6 (24.1) | 76.1 (25.8)
  PEDS QOL Psychosocial Health Summary Score | 73.5 (21.6) | 64.4 (19.9)
  PEDS QOL Total Score | 79 (16.4) | 67 (20.4)

6. Primary Outcome: Quality of Life and Social/Emotional Functioning
Description: as for outcome 5
Time Frame: At 12 week follow up after Baseline
Population: Only adolescents under age 18 received the PEDS-QOL measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 19 | 9
score on a scale
  PEDS QOL Physical Score | 87.2 (15.2) | 74 (20.4)
  PEDS QOL Emotional Score | 63.7 (25.4) | 50.6 (20.7)
  PEDS QOL Social Score | 82.6 (27.6) | 72.2 (29.4)
  PEDS QOL Psychosocial Health Summary Score | 72.8 (23.2) | 61.7 (16.4)
  PEDS QOL Total Score | 77.8 (19.3) | 65.9 (16.4)

7. Primary Outcome: Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication)
Description: The Child and Adolescent Service Assessment (CASA) collects service utilization of all participants to determine the amount of services accessed. The CASA response data displayed are those who responded positively that they received the service. Those who said yes to receiving the service is scored as a 1. Multiple participants can say yes to more than 1 service.
Time Frame: 4 week follow up
Population: 6 intervention participants did not complete week 4 assessment and 1 TAU participant did not complete week 4 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 62 | 32
Participants
  Use outpatient services | 45 | 25
  Use school services | 5 | 2
  Use emergency services | 0 | 0
  Use legal services | 0 | 0
  Use inpatient services | 1 | 0
  Use medications | 33 | 18

8. Primary Outcome: Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication)
Description: as for outcome 7
Time Frame: 12 week follow up
Population: 9 intervention participants did not complete week 12 assessment and 2 TAU participants did not complete week 12 assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath | Treatment As Usual (TAU)
Number analyzed (Participants) | 59 | 31
Participants
  Use outpatient services | 45 | 23
  Use school services | 4 | 1
  Use emergency services | 0 | 0
  Use legal services | 0 | 0
  Use inpatient services | 1 | 0
  Use medications | 32 | 14

9. Secondary Outcome: Application Utilization-BRITE App Use by Participants
Description: Use of the technical components of interventions and web portals for BRITEPath with be monitored throughout Phase 2. Utilization will be measured by the number of participants who have engaged with the application over time, including rating distress levels in the app and utilizing the following app features: learn to savor, reaching out to contacts, soothe breathe, sooth guided meditation, crisis survival strategies, distract with happy thoughts, distract exercise, savor, and soothe activities to help you sleep.
Time Frame: Up to 12 week follow up
Population: 68/68 participants received the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 68
Participants
  First distress level: Completed | 37
  First distress level: Did not complete | 31
  Second distress level: Completed | 29
  Second distress level: Did not complete | 39
  Learn to savor: Completed | 4
  Learn to savor: Did not complete | 64
  Reaching out to contacts: Completed | 11
  Reaching out to contacts: Did not complete | 57
  Soothe Breathe: Completed | 17
  Soothe Breathe: Did not complete | 51
  Soothe Guided Meditation: Completed | 9
  Soothe Guided Meditation: Did not complete | 59
  Crisis survival strategies: Completed | 14
  Crisis survival strategies: Did not complete | 54
  Distract with happy thoughts: Completed | 17
  Distract with happy thoughts: Did not complete | 51
  Distract exercise: Completed | 13
  Distract exercise: Did not complete | 55
  Savor: Completed | 15
  Savor: Did not complete | 53
  Soothe activities to help you sleep: Completed | 10
  Soothe activities to help you sleep: Did not complete | 58

10. Secondary Outcome: Application Utilization-Number of Participants With Provider Who Completed Guide2BRITE Onboarding Process
Description: Use of the technical components of interventions and web portals for BRITEPath with be monitored throughout Phase 2. Use of the technical components of Guide2BRITE and the BRITEPortal for physicians will be monitored throughout Phase 1b. Utilization will be measured by the number of providers who have completed the Guide2BRITE onboarding process which includes steps 1, 1.2, 1.3, 2, 2.1, 2.2, 2.3, 2.4, 2.5, 3, 3.2, 4, 4.1, and 5. Each step includes text field components of a standard safety plan that needs to be completed. Providers who clicked "next" at each step after filling in the text boxes were counted.
Time Frame: Up to 12 week follow up
Population: 68/68 participants were onboarded by clinician.
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 68
Participants
  Step 1: Completed | 41
  Step 1: Did not complete | 27
  Step 1.2: Completed | 41
  Step 1.2: Did not complete | 27
  Step 1.3: Completed | 41
  Step 1.3: Did not complete | 27
  Step 2: Completed | 0
  Step 2: Did not complete | 68
  Step 2.1: Completed | 41
  Step 2.1: Did not complete | 27
  Step 2.2: Completed | 41
  Step 2.2: Did not complete | 27
  Step 2.3: Completed | 41
  Step 2.3: Did not complete | 27
  Step 2.4: Completed | 41
  Step 2.4: Did not complete | 27
  Step 2.5: Completed | 41
  Step 2.5: Did not complete | 27
  Step 3: Completed | 41
  Step 3: Did not complete | 27
  Step 3.2: Completed | 41
  Step 3.2: Did not complete | 27
  Step 4: Completed | 0
  Step 4: Did not complete | 68
  Step 4.1: Completed | 40
  Step 4.1: Did not complete | 28
  Step 5: Completed | 2
  Step 5: Did not complete | 66

11. Secondary Outcome: Cost Estimate for Implementation of BRITEPath Intervention
Description: An overall average of the cost of implementing the BRITEPath intervention (including labor, equipment, supplies, facilities) will be estimated. Outcome measure data below highlights the estimated cost of the intervention BRITEPath Intervention per participant, measures were based on estimates from staff and not on empirical data at the individual level.
Time Frame: At 12 week follow up after Baseline
Population: 68/68 participants received BRITEPath onboarding
Measure: Mean (Full Range); unit: dollars per participant
Arm/Group | BRITEPath
Number analyzed (Participants) | 68
dollars per participant | 457.43 [214.10 to 597.05]

12. Secondary Outcome: Usability and Satisfaction
Description: Satisfaction to BRITEPath will be assessed through questions developed by investigators to understand experience with the program. Questions investigators have adapted from literature reviews on satisfaction include: "If a friend were in need of mental health care for depression or suicidal thoughts or behaviors, would you recommend BRITEPath to help him/her manage symptoms?" The response options include: No, definitely not; No, I don't think so; Yes, I think so; Yes, definitely
Time Frame: At exit interview following week 4 study visit or week 12 study visit (depending on when youth attends mental health session that uses BRITEPath tools)
Population: 51 participants responded to 2 of the exit interview items and 50 participants responded to the 3rd exit interview item
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 51
Participants
  No, definitely not | 8
  No don't think so | 8
  Yes, I think so | 19
  Yes, definitely | 16

13. Secondary Outcome: Usability and Satisfaction
Description: Satisfaction to BRITEPath will be assessed through questions developed by investigators to understand experience with the program. Questions investigators have adapted from literature reviews on satisfaction include: "How satisfied are you with the amount of help you received?" The response options include: Very Dissatisfied, Dissatisfied, Satisfied, Very Satisfied
Time Frame: as for outcome 12
Population: 51 participants responded to 2 of the exit interview items and 50 participants responded to the 3rd exit interview item
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 51
Participants
  Very Dissatisfied | 5
  Dissatisfied | 6
  Satisfied | 30
  Very Satisfied | 10

14. Secondary Outcome: Usability and Satisfaction
Description: Satisfaction to BRITEPath will be assessed through questions developed by investigators to understand experience with the program. Questions investigators have adapted from literature reviews on satisfaction include: "Have the services you received helped you to deal more effectively with your problem?" The response options include: Seemed to make things worse, Really didn't help, Yes, somewhat, or Yes, a great deal.
Time Frame: as for outcome 12
Population: 51 participants responded to 2 of the exit interview items and 50 participants responded to the 3rd exit interview item
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 50
Participants
  Seemed to make things worse | 2
  Really didn't help | 11
  Yes, somewhat | 26
  Yes, a great deal | 11

15. Secondary Outcome: Satisfaction With Technical Components
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ). The PSSUQ is 19 items with response options ranging from 1 to 7 where 1= strongly disagree and 7= strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. Questions from sub-domains were chosen to tailor the questioning to this particular intervention.
Time Frame: as for outcome 12
Population: Some participants did not respond to all questions in PSSUQ measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath
Number analyzed (Participants) | 51
score on a scale
  Overall, I am satisfied with how easy it is to use BRITE App.: number analyzed (Participants) | 50
  Overall, I am satisfied with how easy it is to use BRITE App. | 4.7 (2)
  The information provided with BRITE App such as online help was clear: number analyzed (Participants) | 40
  The information provided with BRITE App such as online help was clear | 5.2 (2.1)
  The information provided with BRITE App such as notifications to rate my mood was clear: number analyzed (Participants) | 40
  The information provided with BRITE App such as notifications to rate my mood was clear | 5 (2.1)
  The information provided during the onboarding with my therapist was clear: number analyzed (Participants) | 40
  The information provided during the onboarding with my therapist was clear | 5.3 (2)
  I liked interacting with the BRITE app program: number analyzed (Participants) | 50
  I liked interacting with the BRITE app program | 4.6 (1.9)
  I needed to learn a lot of things before I could get going with BRITE App | 1.8 (1.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over course of open enrollment and follow up data collection (11/05/2020 to 03/23/2022). Adverse event data was collected for each individual over 12 weeks that they were engaged in the study.
Arm/Group | BRITEPath | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/33
Other Adverse Events (participants affected / at risk) | 1/68 | 0/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRITEPath (N=68) | Treatment As Usual (TAU) (N=33)
Unanticipated problem-Breach of confidentiality (Psychiatric disorders) | 1 (1) | 0 (0) — Patient name was inadvertently sent to wrong study practice when they were randomized to intervention. Research staff notified the IRB and they felt no additional reporting was necessary and was unrelated to study intervention.

LIMITATIONS AND CAVEATS:
The small sample size of this pilot study was selected for feasibility testing, not for hypothesis testing; thus, inferential tests were underpowered and conducted for exploratory purposes. It lacked a full control group we originally intended to collect. The impact of treatment on individuals who dropped out of treatment and on those lost during follow-up is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT04672798/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04672798/ICF_002.pdf